CLINICAL TRIAL: NCT06855979
Title: The Impact of Dietary Intervention Using Innovative Food with High Antioxidant Potential on Oxidative/antioxidant Markers in Blood and Gut Microbiota in Athletes
Brief Title: The Impact of Dietary Intervention on Oxidative/antioxidant Markers and Gut Microbiota in Athletes
Acronym: SportDiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APK.002.405.2024; SKN/SP/601112/2024 (Other Grant/Funding Number: Ministry of Science and Higher Education in Poland); B.SUB.25.207 (Other Grant/Funding Number: Medical University of Bialystok)
Record Dates: First submitted 2025-02-20; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Non Communicable Diseases
Keywords: sport; cardiovascular disease; antioxidant stress
MeSH Terms: conditions — Noncommunicable Diseases; Cardiovascular Diseases | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxidative-antioxidant markers in blood and gut microbiota (Experimental): Before and after the 1-month dietary intervention, the following markers will be determined in the blood: antioxidant potential, antioxidant enzymes, oxidative stress. Moreover, the intestinal microbiota will be determined before and after the intervention.
  Interventions: Other: Food with high antioxidant potential

INTERVENTIONS:
Other: Food with high antioxidant potential — The dietary intervention using fruit and nut bars with high antioxidant activity will last 1 month. Before and after the procedure, oxidative-antioxidant markers in the blood and intestinal microflora in the stool will be determined.

SUMMARY:
During intense physical exercise, there is an overproduction of reactive oxygen species, which leads to oxidative stress and reduced training and sports performance, as well as the development of chronic diseases. Eating foods with a high content of bioactive ingredients and high antioxidant potential can alleviate the negative effects caused by reactive oxygen species and improve the state of intestinal microflora.

The aim of these interventional studies was to determine whether daily consumption of foods with high antioxidant potential, including fruit and nut bars, for a period of 1 month would reduce oxidative stress in athletes during competition and positively change the intestinal microflora.

DETAILED DESCRIPTION:
The study concerns a 4-week dietary intervention. The intervention consisted of daily consumption of 1 bar weighing 50 g, containing nuts and dried fruits with high antioxidant potential. The study included a group of 50 women and men, healthy athletes (cyclists, long-distance runners and triathletes). A 3-day, 24-hour dietary interview was conducted before and after the dietary intervention. Then, using the Dieta 6.0 computer program, the energy and nutrient contents in the diet were estimated. In addition, adherence to the dietary intervention was assessed using a survey questionnaire. Before and after the dietary intervention, oxidative-antioxidant markers were determined in the blood of the subjects (oxidative stress, antioxidant potential, concentration of antioxidant enzymes: glutathione peroxidase, superoxide dismutase, catalase) using ready-made kits. Moreover, changes in the intestinal microbiome were assessed in feces before and after the dietary intervention. Additionally, height and weight were measured before and after the intervention to calculate body mass index (BMI). The study will help answer the question of whether dietary intervention using foods with high antioxidant potential can influence changes in oxidative-antioxidant markers in the blood, intestinal microbiome and body weight of study participants.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women with high physical activity (triathletes, cyclists, long-distance runners), not taking medications for chronic diseases, age 20-50 years, men and women.

Exclusion Criteria:

* occurence of chronic diseases (e.g. hypertension, diabetes, cancer, thyroid diseases, neurodegenerative diseases), taking medications for chronic diseases, age<20 and >50 years, low physical activity

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Change in antioxidant potential after dietary intervention | 4 weeks
  Before and after the dietary intervention, the antioxidant potential in the blood was determined using the ABTS method.
Change in gut microbiota after dietary intervention | 4 weeks
  The gut microbiota in feces was determined before and after the dietary intervention in a hospital laboratory.
Assessment of dietary intervention | 4 weeks
  The dietary intervention lasted 4 weeks. The subjects received one bar a day weighing 50 g, containing nuts and dried fruits with high antioxidant potential and high polyphenol content. After the dietary intervention, the participants completed a survey containing questions about compliance with the recommendations of the dietary intervention.
Change in blood glutathione peroxidase concentration after dietary intervention | 4 weeks
  Before and after the dietary intervention, the concentration of glutathione peroxidase enzyme in blood was assessed using ready-made laboratory kits.
Change in superoxide dismutase concentration after dietary intervention | 4 weeks
  Before and after the dietary intervention, the concentration of superoxide dismutase enzyme in blood was assessed using ready-made laboratory kits.
Change in catalase concentrations after dietary intervention | 4 weeks
  Before and after the dietary intervention, the concentration of catalase enzyme in blood was assessed using ready-made laboratory kits.
Change in oxidative stress after dietary intervention | 4 weeks
  Before and after the dietary intervention, the oxidative stress in blood was assessed using ready-made laboratory kits.

SECONDARY OUTCOMES:
Assessment of dietary nutrients before and after dietary intervention | 4 weeks
  Before and after the dietary intervention, a 3-day, 24-hour interview was conducted regarding the consumption of products and dishes during the day. Using the Diet 6.0 computer program, the content of individual nutrients in the diet and energy of diet were determined.
Body weight assessment before and after dietary intervention | 4 weeks
  The change in body weight of the subjects before and after the dietary intervention was determined using a scale in kilograms with an accuracy of 100 g.
Measuring the height of study participants | 4 weeks
  Height was determined in centimeters using a measuring tape with an accuracy of 1 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata E Zujko, Prof., Principal Investigator — Medical University of Bialystok, Jana Kilinskiego 1, 15-089 Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
The research results will be published in a scientific journal. Detailed data of respondents are not made available due to personal data protection.
Supporting Information: CSR
Time Frame: The clinical trial report will be published in scientific journals after the study is completed.
Access Criteria: Additional information can be obtained by writing to the principal investigator's address: malgorzata.zujko@umb.edu.pl.